CLINICAL TRIAL: NCT02800525
Title: The Comparison of Picosecond 532 and 1,064 Nanometers Laser and Q-switched Nd:YAG 532 and 1,064 Nanometers Laser in the Treatment of Benign Pigmented Lesions: A Randomized Controlled Trial
Brief Title: Comparison of Picosecond and Q-switched Laser for Benign Pigmented Lesions Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Si468/2016 (EC1)
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-06

CONDITIONS: Benign Pigmented Lesions
Keywords: Benign pigmented lesions; Picosecond laser; Q-switched laser

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Picosecond laser (Experimental): The pigmented lesions on this half-side of the face would be treated with picosecond laser.
  For epidermal lesions, 1 laser treatment would be performed. For dermal lesions, 5 laser treatments would be performed every 3 month-interval.
  The wavelength of 532 or 1064 nm would be chosen for appropriate lesions
  Interventions: Device: Picosecond laser
- Q-switched Nd:YAG laser (Active Comparator): The pigmented lesions on this half-side of the face would be treated with q-switched Nd:YAG laser.
  For epidermal lesions, 1 laser treatment would be performed. For dermal lesions, 5 laser treatments would be performed every 3 month-interval.
  The wavelength of 532 or 1064 nm would be chosen for appropriate lesions
  Interventions: Device: Q-switched Nd:YAG laser

INTERVENTIONS:
Device: Picosecond laser — Picosecond 532 and 1064 nm laser Treatment of facial pigmented lesions. The energy using depends on the endpoint of immediate whitening of the lesions. The wavelength using depends on the depth of lesions.
  Arms: Picosecond laser
Device: Q-switched Nd:YAG laser — Q-switched Nd-YAG 532 and 1064 nm laser. Treatment of facial pigmented lesions. The energy using depends on the endpoint of immediate whitening of the lesions. The wavelength using depends on the depth of lesion.
  Arms: Q-switched Nd:YAG laser

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of picosecond 532 and 1,064 nanometers laser in the treatment of benign pigmented lesions compared with q-switched 532 and 1,064 nanometers laser.

DETAILED DESCRIPTION:
Benign pigmented lesions can be divided into epidermal lesions such as freckles, lentigines, solar lentigines or cafe au lait macules and dermal lesions such as Nevus of Ota or Hori's nevus.

Q-switched 532 and 1064 nm lasers were reported to be safe and effective in the treatment of these benign pigmented lesions. By using selective photothermolysis theory, both q-switched 532 and 1064 nm lasers target on melanin causes photomechanical destruction of the melanin. However, the occurrence of post inflammatory hyperpigmentation (PIH) were reported especially in patients with darker skin type.

Recently, picosecond 532, 755, 1064 nm laser was reported to treat benign pigmented lesions effectively. With their ultra short pulse duration (picosecond domain), it is ideally believed to be pure photomechanical effects without thermal injury to surrounding tissue. As a result, the incident of PIH should be reduced.

The investigators then aimed to compared the efficacy and efficacy of different pulse duration between nanosecond and picosecond laser in the treatment of benign pigmented lesions.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* having any benign pigmented lesions on both sides of the face or any tattoo on any part of body which would like to be removed
* Fitzpatrick skin phototype 3-5

Exclusion Criteria:

* Previously treated with any laser within 3 months before enrollment into the study
* Patients with lesions with any clinical suspicion of being pre-cancerous or skin malignancies of any kind
* Patients who have photosensitive dermatoses
* Pregnancy and lactation woman
* Patients with wound infections (herpes, other) on the day of treatment
* Patients with moderate and severe inflammatory acne, Immunosuppressed patients, history of vitiligo
* Patients with unrealistic concerns/expectations and inability to do the appropriate post-operative care

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Doctor evaluation of improvement using quartile scale | For epidermal lesion: 1 and 3 months after 1 laser treatment. For dermal lesion: 1, 3 and 6 months after 5 laser treatments
  Quartile scale 0-4

SECONDARY OUTCOMES:
Side effect occurrence | immediately after treatments, 2, 3, 4, and 12 weeks after the 1st laser treatment, and added more 1, 3 and 6 months after 5 laser treatments for dermal lesions
Patients evaluation of improvement using quartile scale | For epidermal lesion: 1 and 3 months after 1 laser treatment. For dermal lesion: 1, 3 and 6 months after 5 laser treatments

CONTACTS AND LOCATIONS:
Overall Officials: Woraphong Manuskiatti, Prof., M.D., Principal Investigator — Department of Dermatology, Siriraj Hospital
Locations (1):
- Department of Dermatology, Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Result] Friedman DJ. Successful Treatment of a Red and Black Professional Tattoo in Skin Type VI With a Picosecond Dual-Wavelength, Neodymium-Doped Yttrium Aluminium Garnet Laser. Dermatol Surg. 2016 Sep;42(9):1121-3. doi: 10.1097/DSS.0000000000000780. No abstract available. PMID 27227473
- [Result] Levin MK, Ng E, Bae YS, Brauer JA, Geronemus RG. Treatment of pigmentary disorders in patients with skin of color with a novel 755 nm picosecond, Q-switched ruby, and Q-switched Nd:YAG nanosecond lasers: A retrospective photographic review. Lasers Surg Med. 2016 Feb;48(2):181-7. doi: 10.1002/lsm.22454. PMID 26922302
- [Result] Chan JC, Shek SY, Kono T, Yeung CK, Chan HH. A retrospective analysis on the management of pigmented lesions using a picosecond 755-nm alexandrite laser in Asians. Lasers Surg Med. 2016 Jan;48(1):23-9. doi: 10.1002/lsm.22443. Epub 2015 Dec 22. PMID 26696500
- [Result] Bogdan Allemann I, Goldberg DJ. Benign pigmented lesions. Curr Probl Dermatol. 2011;42:81-96. doi: 10.1159/000328267. Epub 2011 Aug 16. PMID 21865801
- [Result] Bukvic Mokos Z, Lipozencic J, Ceovic R, Stulhofer Buzina D, Kostovic K. Laser therapy of pigmented lesions: pro and contra. Acta Dermatovenerol Croat. 2010;18(3):185-9. PMID 20887701